CLINICAL TRIAL: NCT04783324
Title: The Effect of the E-Mobile Health Application for Pregnant Women Created Based on the Roy's Adaptation Model on Postpartum Adaptation
Brief Title: The Effect of the E-Mobile Health Application on Postpartum Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ozkan, Principal investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SultanOzkan
Record Dates: First submitted 2021-01-22; First posted 2021-03-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Postpartum Period; Pregnant Women; Adaptation; Mobile Applications
Keywords: Mobile Applications; Postpartum Period; Adaptation; Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: The study consists of two groups: Experimental group and control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Pregnant women in the intervention group will use the e-mobile health application developed by the researcher.
  Interventions: Behavioral: E-Mobile Health Application
- Control Group (No Intervention): Pregnant women in the control group will not be intervened and standard care will be applied.

INTERVENTIONS:
Behavioral: E-Mobile Health Application — The e-mobile health application prepared by the researcher will be used. E-mobile health application include information about postpartum care.
  Arms: Experimental Group

SUMMARY:
The purpose of this research is to determine the effect of the e-mobile health application on postpartum adaptation. The study will consist of two groups: Experimental group and control group.

DETAILED DESCRIPTION:
This is a randomized controlled trial. A questionnaire and The Postpartum Self-Evaluation Questionnaire will be used to collect data. The main hypothesis of the research: Postpartum Self-Evaluation Questionnaire total mean score of women who use e-mobile health application created according to Roy's Adaptation Model is not different from the total mean score of women in the control group.

Research sample will consist of a total of 62 pregnant women, 31 in the experimental group and 31 in the control group. The data will be evaluated with the SPSS (Statistical Package of SocialSciences) 24.0 package program.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* Being in the 32nd week of pregnancy and above
* Not getting any diagnosis that poses a risk for pregnancy (Multiple pregnancy, Gestational Diabetes, Preeclampsia, Eclampsia, Placenta Previa, Fetal Anomaly, Intrauterine Growth Retardation)
* Speaking Turkish
* To be at least a primary school graduate
* Having a smart phone with Android operating system

Exclusion Criteria:

* Multiparous
* Being under 32 weeks of pregnancy
* Getting any diagnosis that poses a risk to pregnancy (Multiple pregnancy, Gestational Diabetes, Preeclampsia, Eclampsia, Placenta Previa, Fetal Anomaly, Intrauterine Growth Retardation)
* Not speaking Turkish
* Having a smartphone with an operating system other than Android

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Postpartum Adaptation | At postpartum tenth day (baseline) and last-interview at postpartum sixth week (change from baseline at sixth week)
  Postpartum adaptation according to Postpartum Self Evaluation Scale. Postpartum self evaluation questionnaire consists of 82 questions in total. The questions are scored between 1 and 4 points. The minimum value that can be obtained from the scale is 82, the maximum value is 328. It is seen that the lower the score in this scale, the higher the postpartum adaptaion of the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Şengül Yaman Sözbir, PhD, Principal Investigator — Gazi University
Locations (1):
- Ankara Koru Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozkan Sat S, Yaman Sozbir S. Randomized Controlled Trial of a Mobile Health Application Based on Roy's Adaptation Model on Postpartum Adaptation. Nurs Res. 2023 May-Jun 01;72(3):E16-E24. doi: 10.1097/NNR.0000000000000647. Epub 2023 Feb 21. PMID 36920158